CLINICAL TRIAL: NCT04800315
Title: A Phase 2, Multicenter, Global, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Safety and Efficacy of Cendakimab (CC-93538) in Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate Safety and Effectiveness of Cendakimab (CC-93538) in Participants With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-93538-AD-001; 1111-1260-5462 (Registry Identifier: WHO); 2020-005212-22 (EudraCT Number)
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Dermatitis, Atopic; Eczema
Keywords: Atopic Dermatitis; Cendakimab; CC-93538
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — cendakimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose 1: CC-93538 SC QW (Experimental): Administration of CC-93538 Subcutaneous (SC) Once weekly (QW) for 16 weeks.
  Interventions: Drug: CC-93538
- Dose 2: CC-93538 SC Q2W and Placebo alternating every other week SC Q2W (Experimental): Starting at the baseline visit, active IP will be administered. On the alternate weeks, placebo will be administered to maintain the blind.
  Interventions: Drug: CC-93538; Other: Placebo
- Dose 3: CC-93538 SC Q2W and Placebo SC weekly (Experimental): Starting at the baseline visit, active IP and matching placebo will be administered.
  On the alternate weeks, placebo will be administered weekly to maintain the blind.
  Interventions: Drug: CC-93538; Other: Placebo
- Placebo SC QW (Placebo Comparator): Administration of placebo each week.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CC-93538 — Specified dosages on specified days
  Other Names: RPC4064; cendakimab
  Arms: Dose 1: CC-93538 SC QW; Dose 2: CC-93538 SC Q2W and Placebo alternating every other week SC Q2W; Dose 3: CC-93538 SC Q2W and Placebo SC weekly
Other: Placebo — Specified dosages on specified days
  Arms: Dose 2: CC-93538 SC Q2W and Placebo alternating every other week SC Q2W; Dose 3: CC-93538 SC Q2W and Placebo SC weekly; Placebo SC QW

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of 3 dose regimen of CC-93538 in adult participants with moderate to severe Atopic Dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following criteria to be enrolled in the study:

1. Participant must be ≥ 18 years and ≤ 75 years of age and have a body weight of ≥ 40 kg (88.2 lb) at the time of signing the informed consent form (ICF).
2. Participant has chronic atopic dermatitis (AD) as defined by Hanifin and Rajka that has been present for ≥ 1 year prior to the baseline visit (Day 1).
3. Participant has moderate to severe, active, and symptomatic AD defined by meeting all of the following criteria on the day of the baseline visit (Day 1):

   1. Body Surface Area (BSA) ≥ 10%, and
   2. EASI score ≥ 16, and
   3. vIGA-AD ≥ 3, and
   4. Pruritus Numeric Rating Scale (NRS) severity score ≥ 4.
4. Participant must have a documented history of inadequate response to treatment with topical medications for at least 4 weeks, unless topical treatments are otherwise medically inadvisable or has required systemic therapy for control of disease.
5. Participant must be willing to apply a stable dose of topical emollient (eg, over-the-counter moisturizer, non-medicated emollient, etc.) twice daily for ≥ 7 days prior to the Baseline visit and continue application throughout the study.
6. Participant must commit to avoid prolonged exposure to the sun and not to use tanning booths, sun lamps or other ultraviolet light sources during the study.
7. Participants currently receiving concomitant medications for any reason other than AD, such as inhaled corticosteroids, leukotriene receptor antagonists (eg, montelukast), or mast cell stabilizers (eg, cromolyn sodium) for asthma, must be on a stable regimen, which is defined as not starting a new drug, changing, or stopping dosage within 7 days or 5 half-lives (whichever is longer) prior to Day 1 and through the treatment duration of the study.
8. Female participants of childbearing potential must agree to practice a highly effective method of contraception.

Exclusion Criteria:

1. The presence of any of the following will exclude a participant from enrollment: Evidence of an active and/or concurrent inflammatory skin condition (eg, seborrheic dermatitis, psoriasis, acute allergic contact dermatitis, etc.) that would interfere with the Investigator or participant-driven evaluations of AD.
2. Evidence of acute AD flare between the Screening and Baseline/ Randomization (eg, doubling of the EASI score between Screening and Baseline).
3. Use of topical treatments that could affect the assessment of AD (eg, corticosteroids, calcineurin inhibitors, tars, antibiotic creams, topical antihistamines) within 7 days of the Day 1 visit.
4. Received phototherapy narrowband UVB (NB-UVB) or broad band phototherapy within 4 weeks prior to the Baseline visit.
5. Evidence of immunosuppression, participant is receiving, or has received systemic immunosuppressive or immunomodulating drugs (eg, azathioprine, cyclosporine, systemic corticosteroids, interferon gamma (IFN-γ), Janus kinase inhibitors, methotrexate, mycophenolate-mofetil, etc.) within 4 weeks prior to the Baseline visit.
6. Treatment with immunomodulatory biologics
7. Concurrent treatment with another IP
8. Received a live attenuated vaccine within 1 month prior to the first Screening Visit or anticipates the need to be vaccinated with a live attenuated vaccine during the study.
9. Active parasitic/helminthic infection or a suspected parasitic/helminthic infection.
10. Ongoing infection
11. A history of idiopathic anaphylaxis or a major immunologic reaction (such as anaphylactic reaction, anaphylactoid reaction, or serum sickness) to an immunoglobulin G (IgG) containing agent. A known hypersensitivity to any ingredient in the investigational product (IP) is also exclusionary.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (157):
- United States (62):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Local Institution - 119, Birmingham, Alabama
  - Cahaba Dermatology, Birmingham, Alabama
  - Local Institution - 114, Birmingham, Alabama
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Local Institution - 129, Hot Springs, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Local Institution - 105, Fountain Valley, California
  - George Washington University School of Medicine and Health Sciences, Washington D.C., District of Columbia
  - Local Institution - 128, Washington D.C., District of Columbia
  - Total Vein and Skin, LLC, Boynton Beach, Florida
  - Local Institution - 106, Delray Beach, Florida
  - Palm Beach Dermatology Group, Delray Beach, Florida
  - GCP Global Clinical Professionals, St. Petersburg, Florida
  - Local Institution - 135, St. Petersburg, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Local Institution - 101, Tampa, Florida
  - Local Institution - 103, West Palm Beach, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Aeroallergy Research Labs of Savannah, Savannah, Georgia
  - Local Institution - 134, Savannah, Georgia
  - Local Institution - 108, Springfield, Illinois
  - Sneeze Wheeze and Itch Associates LLC, Springfield, Illinois
  - DS Research, Clarksville, Indiana
  - Local Institution - 115, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Local Institution - 110, Indianapolis, Indiana
  - Local Institution - 107, West Lafayette, Indiana
  - Randall Dermatology, West Lafayette, Indiana
  - Local Institution - 138, Westfield, Indiana
  - Randall Dermatology - Westfield Campus, Westfield, Indiana
  - Kansas City Dermatology P.A., Overland Park, Kansas
  - Local Institution - 116, Overland Park, Kansas
  - DS Research, Louisville, Kentucky
  - Local Institution - 117, Louisville, Kentucky
  - DermAssociates, Silver Spring, Maryland
  - Local Institution - 125, Silver Spring, Maryland
  - Local Institution - 133, Clarkston, Michigan
  - Skin Research Clarkston/Clarkston Dermatology, Clarkston, Michigan
  - Local Institution - 137, Omaha, Nebraska
  - Skin Specialists PC, Omaha, Nebraska
  - JDR Dermatology Research, LLC, Las Vegas, Nevada
  - Local Institution - 121, Las Vegas, Nevada
  - Local Institution - 112, Hackensack, New Jersey
  - Skin Laser and Surgery Specialists of New York and New Jersey LLC, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, Great Neck, New York
  - Local Institution - 130, Great Neck, New York
  - Local Institution - 126, New York, New York
  - Sadick Research Group, New York, New York
  - Central Sooner Research, Norman, Oklahoma
  - Local Institution - 111, Norman, Oklahoma
  - Local Institution - 127, Tulsa, Oklahoma
  - Vital Prospects Clinical Research Institute PC - CRN - PPDS, Tulsa, Oklahoma
  - Local Institution - 109, Portland, Oregon
  - Oregon Medical Research Center, P.C., Portland, Oregon
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Local Institution - 123, Johnston, Rhode Island
  - International Clinical Research, Murfreesboro, Tennessee
  - Local Institution - 100, Murfreesboro, Tennessee
  - Clinical Research Partners LLC, Henrico, Virginia
  - Local Institution - 104, Richmond, Virginia
  - West End Dermatology Associates, Richmond, Virginia
- Canada (18):
  - Institute for Skin Advancement, Calgary, Alberta
  - Local Institution - 203, Calgary, Alberta
  - Local Institution - 213, Edmonton, Alberta
  - Rao Dermatology, Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Local Institution - 207, Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Local Institution - 200, Surrey, British Columbia
  - Local Institution - 205, Winnipeg, Manitoba
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Local Institution - 208, Markham, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - DermEdge, Mississauga, Ontario
  - Local Institution - 211, Mississauga, Ontario
  - Local Institution - 209, Oakville, Ontario
  - The Centre for Clinical Trials Inc., Oakville, Ontario
  - Centre de Recherche Dermatologique du Quebec Metropolitain CRDQ, Québec
  - Local Institution - 202, Québec
- China (4):
  - Kawashima Dermatology, Ichikawa
  - Local Institution - 503, Ichikawa
  - Local Institution - 507, Matsudo
  - Miyata Dermatology Clinic, Matsudo
- Czechia (16):
  - Kozni ambulance Kutna Hora, Kutná Hora
  - Local Institution - 407, Kutná Hora
  - Dermamedica, Náchod
  - Local Institution - 403, Náchod
  - CCBR Ostrava, Ostrava
  - Local Institution - 404, Ostrava
  - Center for Clinical and Basic Research Czech Pardubice, Pardubice
  - Local Institution - 405, Pardubice
  - Clintrial, Prague
  - Local Institution - 402, Prague
  - CCBR Czech Prague s.r.o., Prague
  - Local Institution - 400, Prague
  - FN Motol, Prague
  - Local Institution - 401, Prague
  - Dermatologicka Ambulance MUDr. Petr Trestik, Svitavy
  - Local Institution - 406, Svitavy
- Japan (30):
  - Local Institution - 514, Fukuoka
  - Kyushu Central Hospital of the Mutual Aid Association of Public School Teachers, Fukuoka
  - Local Institution - 504, Fukuoka
  - Fukuoka University Hospital, Fukuoka-shi, Fukuoka
  - Ichinomiya Municipal Hospital, Ichinomiya
  - Local Institution - 506, Ichinomiya
  - Teikyo University Hospital, Itabashi-ku
  - Local Institution - 511, Itabashi-ku
  - Local Institution - 515, Kagoshima
  - Saruwatari Dermatology Clinic, Kagoshima
  - Local Institution - 513, Kofu
  - Yamanashi Prefectual Central Hospital, Kofu
  - Local Institution - 505, Kyoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Charme-Clinique, Matsudo
  - Local Institution - 510, Matsudo
  - Local Institution - 508, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Local Institution - 512, Obihiro
  - Takagi Dermatology, Obihiro
  - Local Institution - 517, Osaka
  - Nakatsu Hifuka Clinic, Osaka
  - Local Institution - 501, Sapporo
  - Medical Corporation Kojinkai Housui Sogo Medical Clinic, Sapporo
  - Local Institution - 500, Sapporo-shi, Hokkaido
  - Sapporo Skin Clinic, Sapporo-shi, Hokkaido
  - Local Institution - 502, Shinjuku
  - Tokyo Medical University Hospital, Shinjuku
  - Local Institution - 509, Yokohoma City, Kanagawa
  - Nomura Dermatology Clinic, Yokohoma City, Kanagawa
- Poland (27):
  - Copernicus Podmiot Leczniczy Sp. z o.o., Gdansk
  - Local Institution - 310, Gdansk
  - Care Clinic, Katowice
  - Local Institution - 309, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Local Institution - 306, Katowice
  - Local Institution - 303, Lodz
  - Specjalistyczne Gabinety Lekarskie DERMED, Lodz
  - Centrum Medyczne Dermoklinika, Lodz
  - Local Institution - 311, Lodz
  - Local Institution - 312, Olsztyn
  - Miejski Szpital Zespolony w Olsztynie, Olsztyn
  - Klinika Zdybski, Ostrowiec Świętokrzyski
  - Local Institution - 300, Ostrowiec Świętokrzyski
  - Laser Clinic Dermatologia Laserowa Medycyna Estetyczna, Szczecin
  - Local Institution - 308, Szczecin
  - Local Institution - 302, Szczecin
  - Twoja Przychodnia Szczecinskie Centrum Medyczne, Szczecin
  - High-Med Przychodnia Specjalistyczna, Warsaw
  - Local Institution - 301, Warsaw
  - Klinika Ambroziak Estederm, Warsaw
  - Local Institution - 307, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
  - Kliniczny Szpital Wojewódzki nr 1 im. F. Chopina w Rzeszowie, Wroclaw
  - Local Institution - 304, Wroclaw
  - Centrum Zdrowia WroMedica, Wroclaw
  - Local Institution - 305, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- [Derived] Blauvelt A, Guttman-Yassky E, Lynde C, Khattri S, Schlessinger J, Imafuku S, Tada Y, Morita A, Wiseman M, Kwiek B, Machkova M, Zhang P, Linaberry M, Li J, Zhang S, Franchin G, Charles ED, De Oliveira CHMC, Silverberg JI. Cendakimab in Patients With Moderate to Severe Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2024 Aug 1;160(8):856-864. doi: 10.1001/jamadermatol.2024.2131. PMID 39018038
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 221 participants Randomized, 220 Participants Treated
Groups:
- Treatment 1: CC-93538 High Dose QW
- Treatment 2: CC-93538 High Dose Q2W
- Treatment 3: CC-93538 Low Dose Q2W
- Placebo: Placebo
Period: Randomization
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Started | 55 | 55 | 55 | 56
Completed (Completed = All randomized participants who recieved at least one dose of study treatment.) | 54 | 55 | 55 | 56
Not Completed | 1 | 0 | 0 | 0
Not completed — Did not receive study treatment | 1 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Started | 54 | 55 | 55 | 56
Completed | 49 | 50 | 52 | 44
Not Completed | 5 | 5 | 3 | 12
Not completed — Adverse Event | 4 | 2 | 1 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 1 | 2 | 2
Not completed — Withdrawal by participant | 0 | 0 | 0 | 4
Not completed — Other Reasons | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo | Total
Number analyzed (Participants) | 55 | 55 | 55 | 56 | 221
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 52 | 51 | 53 | 209
  >=65 years | 2 | 3 | 4 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 26 | 29 | 21 | 95
  Male | 36 | 29 | 26 | 35 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3 | 6
  Not Hispanic or Latino | 53 | 53 | 55 | 53 | 214
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 19 | 14 | 14 | 13 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 8 | 5 | 6 | 23
  White | 30 | 33 | 36 | 37 | 136
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
modified Intent to treat population (mITT) [Count of Participants; unit: Participants] — All enrolled subjects who received at least 1 dose of CC-93538. Same as the safety population.
  Participants | 54 | 55 | 55 | 56 | 220

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change From Baseline in EASI at Week 16
Description: The Eczema Area and Severity Index (EASI) is a composite scoring system assessed by the Investigator based on the proportion of each of the 4 body regions (head and neck, upper limbs, lower limbs, and trunk) affected with Atopic Dermatitis (AD) and the intensity of each of 4 main signs of AD (eg, erythema, induration/papulation, excoriation, and lichenification) and is based on a 4-point scale of 0 (none), 1 (mild), 2 (moderate), and 3 (severe). The sum of the scores is totaled (0 to 72), the lower the score the better.
Time Frame: From initial EASI measurement to week 16
Population: Modified Intent to Treat (mITT) Population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Number analyzed (Participants) | 54 | 55 | 55 | 56
Percent Change | -84.41 (5.07) | -76.03 (4.20) | -78.93 (4.53) | -62.65 (5.53)
Statistical Analysis 1: Comparison: Treatment 1 vs Placebo; Test type: Superiority; p = 0.003, ANCOVA; Mean Difference (Final Values) = -21.76, 95% CI 2-sided [-35.81 to -7.70]
Statistical Analysis 2: Comparison: Treatment 2 vs Placebo; Test type: Superiority; p = 0.057, ANCOVA; Mean Difference (Final Values) = -13.38, 95% CI 2-sided [-27.19 to 0.43]
Statistical Analysis 3: Comparison: Treatment 3 vs Placebo; Test type: Superiority; p = 0.029, ANCOVA; Mean Difference (Final Values) = -16.28, 95% CI 2-sided [-30.88 to -1.68]

2. Secondary Outcome: Percentage of Responders With an vIGA-AD Score of 0 (Clear) or 1 (Almost Clear) and a Reduction ≥ 2 Points From Baseline at Week 16
Description: The Validated Investigator Global Assessment (vIGA-AD) is a validated 5-point assessment intended to assess the global severities of key acute clinical signs of AD, including erythema, induration/papulation, oozing/crusting (lichenification excluded). The rating of clear (0), almost clear (1), mild (2), moderate (3) and severe (4), will be assessed at scheduled visits. The vIGA-AD must be conducted before the EASI assessment. The vIGA-AD is a static evaluation conducted without regard to the score obtained at a previous visit.
  Percentage of responders calculated using Multiple Imputation (MI) approach.
  For participants discontinued study drug, whose vIGA-AD response at Week 16 are missing or cannot be adequately determined (including missing due to COVID-19) without use of rescue therapy/prohibited medication prior to Week 16, their outcomes will be handled using a MI approach assuming missing at random (MAR).
Time Frame: From initial vIGA-AD assessment to week 16
Population: Modified Intent to Treat (mITT) Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Number analyzed (Participants) | 54 | 55 | 55 | 56
Percentage of Participants | 33.3 | 24.4 | 38.2 | 9.4
Statistical Analysis 1: Comparison: Treatment 1 vs Placebo; Test type: Other — Risk Difference; p = 0.004, Cochran-Mantel-Haenszel; Risk Difference VS Placebo = 24.0, 95% CI 2-sided [8.8 to 39.2]
Statistical Analysis 2: Comparison: Treatment 2 vs Placebo; Test type: Other — Risk Difference; p = 0.061, Cochran-Mantel-Haenszel; Risk Difference VS Placebo = 15.3, 95% CI 2-sided [0.8 to 29.8]
Statistical Analysis 3: Comparison: Treatment 3 vs Placebo; Test type: Other — Risk Difference; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference VS Placebo = 28.9, 95% CI 2-sided [13.6 to 44.2]

3. Secondary Outcome: Percentage of EASI-75 Responders at Week 16
Description: The EASI is a composite scoring system assessed by the Investigator based on the proportion of each of the 4 body regions (head and neck, upper limbs, lower limbs, and trunk) affected with AD and the intensity of each of 4 main signs of AD (eg, erythema, induration/papulation, excoriation, and lichenification) and is based on a 4-point scale of 0 (none), 1 (mild), 2 (moderate), and 3 (severe). The sum of the scores is totaled (0 to 72), the lower the score the better.
  Percentage of responders calculated using Multiple Imputation (MI) approach.
  For participants discontinued study drug, whose EASI-75 response at Week 16 are missing or cannot be adequately determined (including missing due to COVID-19) without use of rescue therapy/prohibited medication prior to Week 16, their outcomes will be handled using a MI approach assuming missing at random (MAR).
Time Frame: From initial EASI measurement to week 16
Population: modified Intent to Treat (mITT) population
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Number analyzed (Participants) | 54 | 55 | 55 | 56
Percentage of Participants | 50.0 | 48.2 | 52.7 | 26.3
Statistical Analysis 1: Comparison: Treatment 1 vs Placebo; Test type: Other — Risk Difference; p = 0.018, Cochran-Mantel-Haenszel; Difference VS Placebo = 23.7, 95% CI 2-sided [6.2 to 41.2]
Statistical Analysis 2: Comparison: Treatment 2 vs Placebo; Test type: Other — Risk Difference; p = 0.033, Cochran-Mantel-Haenszel; Difference VS Placebo = 21.8, 95% CI 2-sided [4.3 to 39.3]
Statistical Analysis 3: Comparison: Treatment 3 vs Placebo; Test type: Other — Risk Difference; p = 0.006, Cochran-Mantel-Haenszel; Difference VS Placebo = 26.7, 95% CI 2-sided [9.3 to 44.0]

4. Secondary Outcome: Percentage of EASI-90 Responders at Week 16
Description: The Eczema Area and Severity Index (EASI) is a composite scoring system assessed by the Investigator based on the proportion of each of the 4 body regions (head and neck, upper limbs, lower limbs, and trunk) affected with Atopic Dermatitis (AD) and the intensity of each of 4 main signs of AD (eg, erythema, induration/papulation, excoriation, and lichenification) and is based on a 4-point scale of 0 (none), 1 (mild), 2 (moderate), and 3 (severe). The sum of the scores is totaled (0 to 72), the lower the score the better.
  Percentage of responders calculated using Multiple Imputation (MI) approach.
  For participants discontinued study drug, whose EASI-90 response at Week 16 are missing or cannot be adequately determined (including missing due to COVID-19) without use of rescue therapy/prohibited medication prior to Week 16, their outcomes will be handled using a MI approach assuming missing at random (MAR).
Time Frame: From initial EASI measurement to week 16
Population: Modified Intent to Treat (mITT) Population
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Number analyzed (Participants) | 54 | 55 | 55 | 56
Percentage of participants | 31.5 | 24.0 | 29.1 | 13.4
Statistical Analysis 1: Comparison: Treatment 1 vs Placebo; Test type: Other — Risk Difference; Cochran-Mantel-Haenszel; Risk Difference = 18.1, 95% CI 2-sided [2.3 to 33.9]
Statistical Analysis 2: Comparison: Treatment 2 vs Placebo; Test type: Other — Risk Difference; Cochran-Mantel-Haenszel; Risk Difference = 10.5, 95% CI 2-sided [-4.6 to 25.7]
Statistical Analysis 3: Comparison: Treatment 3 vs Placebo; Test type: Superiority; Cochran-Mantel-Haenszel; Risk Difference = 15.9, 95% CI 2-sided [0.4 to 31.4]

5. Secondary Outcome: Percent Change in Mean SCORAD Scores From Baseline at Week 16
Description: The SCORAD is a validated scoring index for atopic dermatitis, which combines extent (0 to 100), severity (0 to 18), and subjective symptoms (0 to 20) based on pruritus and sleep loss, each scored (0 to 10). The subject will assess the subjective symptoms (itch and sleepless) part of the assessment.
  SCORing Atopic Dermatitis Index (SCORAD) score ranges from 0 to 103, higher scores indicate more severe disease.
Time Frame: From initial SCORAD measurement to week 16
Population: Modified Intent to Treat (mITT) population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Number analyzed (Participants) | 54 | 55 | 55 | 56
Percent Change | -69.28 (4.64) | -55.47 (4.08) | -60.19 (4.38) | -41.11 (5.61)
Statistical Analysis 1: Comparison: Treatment 1 vs Placebo; Test type: Superiority; ANCOVA; Mean Difference (Final Values) = -28.16, 95% CI 2-sided [-41.89 to -14.44]
Statistical Analysis 2: Comparison: Treatment 2 vs Placebo; Test type: Superiority; ANCOVA; Mean Difference (Final Values) = -14.36, 95% CI 2-sided [-27.26 to -1.46]
Statistical Analysis 3: Comparison: Treatment 3 vs Placebo; Test type: Superiority; ANCOVA; Mean Difference (Final Values) = -19.07, 95% CI 2-sided [-33.53 to -4.62]

6. Secondary Outcome: Percent Change From Baseline in Pruritus NRS at Week 16
Description: Pruritus will be assessed by the subject using the Pruritus NRS, which was developed and validated as a single item, patient reported outcome (PRO) of itch severity. Clinical response is indicated by a ≥ 2 to 4-point change from baseline in Peak Pruritus NRS score. The intensity of pruritus will be assessed based on last 24 hours using a validated 11-point NRS, ranging from 0 ("no pruritus") to 10 ("the worst pruritus imaginable").
Time Frame: From initial NRS measurement to week 16
Population: Modified Intent to Treat (mITT) population
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Number analyzed (Participants) | 54 | 55 | 55 | 56
Percent Change | -55.48 (6.22) | -46.15 (5.32) | -49.30 (5.89) | -32.98 (7.46)
Statistical Analysis 1: Comparison: Treatment 1 vs Placebo; Test type: Other — Adjusted Mean Difference VS Placebo; ANCOVA; Adjusted Mean Difference VS Placebo = -22.50, 95% CI 2-sided [-41.46 to -3.54]
Statistical Analysis 2: Comparison: Treatment 2 vs Placebo; Test type: Other — Adjusted Mean Difference VS Placebo; ANCOVA; Adjusted Mean Difference VS Placebo = -13.17, 95% CI 2-sided [-30.67 to 4.33]
Statistical Analysis 3: Comparison: Treatment 3 vs Placebo; Test type: Other — Adjusted Mean Difference VS Placebo; ANCOVA; Adjusted Mean Difference VS Placebo = -16.32, 95% CI 2-sided [-36.40 to 3.75]

7. Secondary Outcome: Percentage of Participants With a Response and Pruritus NRS Change of ≥ 4 Points From Baseline at Week 16
Description: Pruritus will be assessed by the subject using the Pruritus NRS, which was developed and validated as a single item, patient reported outcome (PRO) of itch severity. Clinical response is indicated by a ≥ 2 to 4-point change from baseline in Peak Pruritus NRS score. The intensity of pruritus will be assessed based on last 24 hours using a validated 11-point NRS, ranging from 0 ("no pruritus") to 10 ("the worst pruritus imaginable").
  Percentage of responders calculated using Multiple Imputation (MI) approach.
  For participants discontinued study drug, whose pruritus NRS response at Week 16 are missing or cannot be adequately determined (including missing due to COVID-19) without use of rescue therapy/prohibited medication prior to Week 16, their outcomes will be handled using a MI approach assuming missing at random (MAR).
Time Frame: From initial NRS assessment to week 16
Population: Modified Intent to Treat (mITT) Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Number analyzed (Participants) | 54 | 55 | 55 | 56
Percentage of Participants | 33.3 | 34.5 | 32.7 | 14.8
Statistical Analysis 1: Comparison: Treatment 1 vs Placebo; Test type: Other — Risk Difference VS Placebo; p = 0.042, Cochran-Mantel-Haenszel; Risk Difference VS Placebo = 18.5, 95% CI 2-sided [2.7 to 34.3]
Statistical Analysis 2: Comparison: Treatment 2 vs Placebo; Test type: Other — Risk Difference VS Placebo; p = 0.029, Cochran-Mantel-Haenszel; Risk Difference VS Placebo = 19.9, 95% CI 2-sided [4.1 to 35.7]
Statistical Analysis 3: Comparison: Treatment 3 vs Placebo; Test type: Other — Risk Difference VS Placebo; p = 0.052, Cochran-Mantel-Haenszel; Risk Difference VS Placebo = 18.0, 95% CI 2-sided [2.3 to 33.6]

8. Secondary Outcome: Time to Achieve at Least 4 Points of Improvement in the Severity of Pruritus NRS Scale.
Description: as for outcome 6
Time Frame: From initial NRS pruritus response up to study day 127 (127 days)
Population: Modified Intent to Treat (mITT) Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Number analyzed (Participants) | 54 | 55 | 55 | 56
Days | 54.0 [28.0 to 93.0] | 76.0 [42.0 to 105.0] | 50.0 [27.0 to 111.0] | 123.0 [119.0 to NA] — Not enough events to derive upper limit number via Kaplan-Meier estimates

9. Secondary Outcome: Adjust Mean Percentage Change in BSA in Atopic Dermatitis From Baseline at Week 16
Description: Body Surface Area involvement will be calculated from the sum of the number of handprints of skin afflicted with atopic dermatitis in a body region. The number of handprints of skin afflicted with atopic dermatitis in a body region can be used to determine the extent (%) to which a body region is involved with AD. When measuring, the handprint unit refers to the size of each individual subject's hand with fingers in a closed position. BSA will be calculated by the Investigator or qualified designee using the 1% handprint rule, in which the area represented by the palm with all 5 digits adducted together is approximately 1% of the subject's BSA.
Time Frame: From initial BSA assessment to week 16
Population: Modified Intent to Treat (mITT) Population
Measure: Mean (Standard Error); unit: mean percentage
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Number analyzed (Participants) | 54 | 55 | 55 | 56
mean percentage | -78.85 (6.13) | -64.01 (5.30) | -66.60 (6.03) | -55.73 (6.90)
Statistical Analysis 1: Comparison: Treatment 1 vs Placebo; Test type: Other — Adjusted mean difference VS Placebo; ANCOVA; Adjusted mean difference VS Placebo = -23.12, 95% CI 2-sided [-41.48 to -4.76]
Statistical Analysis 2: Comparison: Treatment 2 vs Placebo; Test type: Other — Adjusted mean difference VS Placebo; ANCOVA; Adjusted mean difference VS Placebo = -8.28, 95% CI 2-sided [-25.16 to 8.59]
Statistical Analysis 3: Comparison: Treatment 3 vs Placebo; Test type: Other — Adjusted mean difference VS Placebo; ANCOVA; Adjusted mean difference VS Placebo = -10.87, 95% CI 2-sided [-29.39 to 7.66]

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment emergent adverse events
Time Frame: From first treatment to the end of follow up, approximately 32 weeks
Population: Modified Intent to Treat (mITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Number analyzed (Participants) | 54 | 55 | 55 | 56
Participants
  Any TEAE | 40 | 41 | 38 | 41
  Any TEAE leading to discontinuation | 4 | 2 | 1 | 2
  Any TEAE of special interest | 9 | 10 | 8 | 10
  Any TESAE | 2 | 1 | 2 | 4

11. Secondary Outcome: Number of Participants With the Presence of Serum Antibodies to CC-93538
Time Frame: From first treatment to the end of follow up, approximately 32 weeks
Population: Modified Intent to Treat (mITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 54 | 55 | 55
Participants
  Baseline ADA Positive | 0 | 3 | 1
  Post Baseline Positive | 22 | 35 | 28
  Post Baseline Negative | 32 | 20 | 27

12. Secondary Outcome: Serum Trough Concentration at Week 16
Description: A serum trough concentration (Ctrough) is the concentration reached by a drug immediately before the next dose is administered. Serum trough concentrations (Ctrough) of CC-93538 will be summarized with descriptive statistics by treatment and visit.
Time Frame: At week 16
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 54 | 55 | 55
ng/mL
  Week 1: number analyzed (Participants) | 51 | 0 | 0
  Week 1 | 66107.2 (31.5) |  |
  Week 2: number analyzed (Participants) | 51 | 52 | 49
  Week 2 | 120157.8 (29.8) | 54957.8 (38.2) | 26651.4 (35.3)
  Week 4: number analyzed (Participants) | 45 | 47 | 48
  Week 4 | 192521.4 (32.8) | 92827.7 (37.6) | 40802.8 (69.8)
  Week 6: number analyzed (Participants) | 47 | 53 | 46
  Week 6 | 220561.6 (55.2) | 108474.6 (48.3) | 43613.1 (99.7)
  Week 8: number analyzed (Participants) | 47 | 48 | 49
  Week 8 | 253107.2 (56.7) | 121185.1 (45.9) | 54975.0 (45.5)
  Week 10: number analyzed (Participants) | 47 | 45 | 47
  Week 10 | 279538.4 (34.9) | 136972.4 (35.6) | 60839.6 (43.6)
  Week 12: number analyzed (Participants) | 45 | 46 | 48
  Week 12 | 310649.1 (36.1) | 137656.3 (40.5) | 57197.5 (104.2)
  Week 14: number analyzed (Participants) | 42 | 51 | 48
  Week 14 | 266531.3 (102.3) | 128517.9 (79.4) | 67212.2 (38.9)
  Week 16: number analyzed (Participants) | 43 | 45 | 55
  Week 16 | 274180.6 (88.0) | 140413.6 (44.0) | 57046.4 (106.8)

13. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Time Frame: From first treatment to the end of follow up, approximately 32 weeks
Population: Modified Intent to Treat Population (mITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
Number analyzed (Participants) | 54 | 55 | 55 | 56
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events (From first treatment to end of study): Approximately 32 Weeks All-Cause mortality (From 1st dose of study to end of study): Approximately 33 Weeks
Description: The number at Risk for All-Cause Mortality represents all treated participants.
  The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/55 | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 2/54 | 1/55 | 2/55 | 4/56
Other Adverse Events (participants affected / at risk) | 34/54 | 35/55 | 29/55 | 34/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=54) | Treatment 2 (N=55) | Treatment 3 (N=55) | Placebo (N=56)
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=54) | Treatment 2 (N=55) | Treatment 3 (N=55) | Placebo (N=56)
Conjunctivitis allergic (Eye disorders) | 4 | 7 | 5 | 2
Fatigue (General disorders) | 3 | 0 | 0 | 1
Injection site erythema (General disorders) | 1 | 0 | 3 | 0
Pyrexia (General disorders) | 0 | 4 | 1 | 5
COVID-19 (Infections and infestations) | 4 | 4 | 3 | 9
Folliculitis (Infections and infestations) | 3 | 2 | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 3 | 2
Respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 5 | 5
Alanine aminotransferase increased (Investigations) | 3 | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 3 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 1
Headache (Nervous system disorders) | 2 | 4 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 20 | 15 | 19 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT04800315/Prot_SAP_000.pdf